CLINICAL TRIAL: NCT01453660
Title: A Pilot Study Measuring Acute Changes in Endothelial Function in Germ Cell Tumor Patients Treated With Cisplatin and Untreated Germ Cell Tumor Controls
Brief Title: Acute Changes in Endothelial Function in Germ Cell Tumor Patients Treated With Cisplatin and Untreated Germ Cell Tumor Controls
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-140
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Germ Cell Cancer
Keywords: Endothelial Function; Endo-PAT2000 system; 11-140
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood, urine

GROUPS / COHORTS (2):
- Cisplatin-Based Chemotherapy Group: GCT patients who are planned to start cisplatin-based chemotherapy will be identified within the genitourinary oncology service clinics and offered inclusion in the trial.
  Interventions: Other: Endo-PAT2000 testing
- Surgery-Only Group: GCT patients who have been treated with surgery and who do not require chemotherapy or radiation will be used as a comparison group to confirm that there is not a significant change in endothelial function among GCT patients treated with surgery alone.
  Interventions: Other: Endo-PAT2000 testing

INTERVENTIONS:
Other: Endo-PAT2000 testing — Endo-PAT2000 testing is done six times during the study. Baseline Assessment Time 1 Cycle 1, Day 1 (Pre-chemotherapy)Time 2 Cycle 1, Day 1 (After 1st dose of cisplatin), Time 3 Cycle 1, Day 2 (Before second cisplatin dose of cycle 1), Time 4 Cycle 1, Day 5 (After last cisplatin dose of cycle 1), End-of-Study Assessment Time 5 (14-34 weeks from Time 1; e.g., 1-12 weeks following completion of the last cycle of first-line chemotherapy) Long-Term Follow Up Assessment Time 6 (24-30 months from Time 1)
  Groups: Cisplatin-Based Chemotherapy Group
Other: Endo-PAT2000 testing — Time 1: A baseline assessment will be performed in the fasting state including Endo-PAT2000, vital signs, waist circumference, fasting blood draw, & urine sample. This will be considered Day 1 of the study for this group of patients. Time 2 (2-5 hours from Time 1): Two to five hours after Time 1, patients will undergo assessment of blood pressure & heart rate, including orthostatics & Endo-PAT2000 testing. Time 5 -- End of Study visit (14-34 weeks from Time 1): At a time point 14 to 34 weeks later than Time 1 patients will undergo study testing in the fasting state. This includes Endo-PAT2000 testing, vital signs including orthostatics, waist circumference, fasting blood draw, & urine sample. The Surgery-Only Group will not have any assessment at Time 3 (Day 2) or Time 4 (Day 5) due to logistical concerns. Long-Term Follow Up Assessment Time 6 (24-30 months following Time 1)
  Other Names: For any patients in Surgery-Only Group who relapse & enroll in the the; Cisplatin-Based Chemotherapy Group before the completion of the Surgery Group; End of Study Assessment, the Baseline Time 1 Chemotherapy Group Assessment can; will also serve as the End of Study Time 5 Surgery Group Assessment.
  Groups: Surgery-Only Group

SUMMARY:
Cisplatin is one of the most common chemotherapy drugs used to treat many different cancers, including germ cell tumors (GCT). Cisplatin is very effective in treating GCT, but there are side effects. One of the possible long-term side effects of cisplatin is thought to be heart disease. The way that cisplatin causes heart disease is not well understood. One possibility is that cisplatin may damage the inside layer of blood vessels called the endothelium. The purpose of this study is to measure changes in the endothelium that happen when patients with GCT get cisplatin chemotherapy and to compare these changes with a group of patients not receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Cisplatin-Based Chemotherapy Group

* Histologically-proven diagnosis of GCT
* Male
* Age ≥18
* No prior exposure to chemotherapy or radiation
* Planned to receive 3-4 cycles of cisplatin-based chemotherapy

Surgery-Only Group

* Histologically-proven diagnosis of GCT Male
* Age ≥18
* Surgical management of GCT performed less than 90 days before start of study (includes orchiectomy and primary retroperitoneal lymph node dissection (RPLND))
* No prior exposure to chemotherapy or radiation

Exclusion Criteria:

Cisplatin-Based Chemotherapy Group

* Prior exposure to chemotherapy or radiation
* Known diagnosis or history of being diagnosed with vasculitis, autonomic dysfunction, coronary artery disease, or collagen-vascular disease

Surgery-Only Group

* Prior exposure to chemotherapy or radiation
* Planned for non-surgical management with chemotherapy or radiation.
* Known diagnosis or history of being diagnosed with vasculitis, autonomic dysfunction, coronary artery disease, or collagen-vascular disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Cisplatin-Based Chemotherapy Group will be recruited from the Genitourinary (GU) oncology clinics. The GU Oncology section has a large clinical service which ensures adequate recruitment.
  The Surgery-Only Group will consist of patients with a diagnosis of GCT who have recently had surgical management of their disease and are not planned to receive radiation or chemotherapy. Potentially eligible patients will be recruited from the GU Oncology and Urology clinics since they are seen by both services.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2011-10-11 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Measure the endothelial reactivity (PAT-RH) in both groups | 15 minutes
  The Endo-PAT quantifies the endothelium-mediated changes in vascular tone, elicited by a 5-minute occlusion of the brachial artery (using a standard BP cuff).

SECONDARY OUTCOMES:
Identify sociodemographic | 2 years
  (age, race/ethnicity)
Identify comorbid health conditions | 2 years
  Other laboratory studies being assessed in this trial will include lipid profile, testosterone, LH, FSH, and hemoglobin A1C. These tests are being evaluated to determine if there are concurrent comorbidities
Measure PAT-RH index | 2 years
  at Time 6 (Long-Term Follow Up Assessment) in the Cisplatin-Based Chemotherapy Group and evaluate long term changes in PATRH index.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Feldman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/3151.cfm